CLINICAL TRIAL: NCT03722498
Title: Randomized Phase Ⅱ Study of Second-line Treatment Comparing Hepatic Arterial Infusion Chemotherapy of Oxaliplatin, 5-fluorouracil and Leucovorin With Sorafenib in Hepatocellular Carcinoma Refractory to Transarterial Chemoembolization
Brief Title: Phase Ⅱ Study of HAIC of FOLFOX vs. Sorafenib in HCC Refractory to TACE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No patients join
Sponsor: Sun Yat-sen University (Other)
Collaborators: Guangzhou No.12 People's Hospital (Other Government); Kaiping Central Hospital (Other)
Responsible Party: Principal Investigator, Shi Ming, Proffesor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC-H171011
Record Dates: First submitted 2018-10-25; First posted 2018-10-29 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatic arterial infusion chemotherapy; Sorafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Oxaliplatin; Fluorouracil; Leucovorin; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HAIC of FOLFOX (Experimental): Hepatic arterial infusion chemotherapy with oxaliplatin, leucovorin, and 5-fluorouracil
  Interventions: Drug: HAIC of FOLFOX
- Sorafenib (Active Comparator): Sorafenib 400 mg orally twice a day
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: HAIC of FOLFOX — administration of oxaliplatin , fluorouracil, and leucovorin via the tumor feeding arteries
  Other Names: Oxaliplatin , fluorouracil, and leucovorin
  Arms: HAIC of FOLFOX
Drug: Sorafenib — administration of Sorafenib
  Arms: Sorafenib

SUMMARY:
To evaluate safety and efficacy of combined hepatic arterial infusion chemotherapy (HAIC) of oxaliplatin, 5-fluorouracil and leucovorin and sorafenib in hepatocellular carcinoma (HCC) refractory to transarterial chemoembolization(TACE)

DETAILED DESCRIPTION:
In most current guidelines, sorafenib is considered as the second-line treatment for patients with transarterial chemoembolization(TACE) failure or refractoriness.However,the median overall survival of those treated with sorafenib monotherapy was 16.4 to 24.7 months.

Whether combining sorafenib with hepatic arterial infusion chemotherapy(HAIC) of oxaliplatin,5-fluorouracil and leucovorin is safe, well tolerated, and efficacious remains unknown, with no prospective clinical data currently available.The investigators therefore conducted a prospective and randomized phase II trial to compare the safety and efficacy of HAIC with sorafenib in patients refractory to TACE

ELIGIBILITY:
Inclusion Criteria:

* TACE failure or refractoriness based on the Liver Cancer Study Group of Japan (LCSGJ) criteria, including appearance of vascular invasion or two or more consecutive insufficient responses of the intrahepatic lesion;
* Except for TACE, patients have received no previous anti-tumor treatment;
* The diagnosis of HCC was based on histological results;
* Patients must have at least one tumor lesion that can be accurately measured;
* Not amendable to surgical resection ,local ablative therapy and any other cured treatment;
* No Cirrhosis or cirrhotic status of Child-Pugh class A only;
* No liver protection therapy in 2 weeks before enrolled, and meet the following laboratory parameters:(a) Platelet count ≥ 75,000/μL; (b)Hemoglobin ≥ 8.5 g/dL;(c) Total bilirubin ≤ 30mmol/L;(d) Serum albumin ≥ 32 g/L;(e) ASL and AST ≤ 5 x upper limit of normal;(f) Serum creatinine ≤ 1.5 x upper limit of normal;(g) INR > 2.3 or PT/APTT within normal limits; (h) Absolute neutrophil count (ANC) >1,500/mm3;
* Ability to understand the protocol and to agree to and sign a written informed consent document

Exclusion Criteria:

* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy;
* Known history of HIV;
* History of organ allograft;
* Known or suspected allergy to the investigational agents or any agent given in association with this trial;
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy;
* Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-03-22 (Estimated); Study Completion 2021-03-22 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 12 months
  The period from the date of the start of HAIC or sorafenib until the date of the confirmation of tumor progression or death

SECONDARY OUTCOMES:
Overall survival | 12 months
  The period from the date of the start of HAIC or sorafenib until the date of the confirmation of tumor progression or death
Adverse Events | 30 Days after HAIC and TACE
  Postoperative adverse events were graded based on CTCAE v4.03
Objective response rate | 12 months
  Best response based on mRECIST

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shi, MD, Principal Investigator — The Department of Hepatobiliary Oncology of Sun Yat-sen University Cancer Center
Locations (3):
- China (3):
  - Guangzhou Twelfth People 's Hospital, Guangzhou, Guangdong
  - Ming Shi, Guangzhou, Guangdong
  - Kaiping Central Hospital, Kaiping, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided